CLINICAL TRIAL: NCT05423314
Title: Participation Rate (Response Rate) and Factors Associated With Non-response to "Online Surveys" in Perioperative Knee Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: "Online Surveys" in Perioperative Knee Anterior Cruciate Ligament (ACL) Reconstruction
Acronym: ORTHENSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: CHU de Toulouse; RnIPH 2021-82 (Other: CHU de Toulouse)
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: patients operated for ACLR
- cold therapy: patients operated for ACLR, and received a "knee brace cold therapy" to use it in the post op recovery rehabilitation, sent to patient's home directly during pre-op phase.
  Interventions: Procedure: knee brace cold therapy

INTERVENTIONS:
Procedure: knee brace cold therapy — receiving a "knee brace cold therapy" to use it in the post op recovery rehabilitation, sent to patient's home directly during pre-op phase.
  Groups: cold therapy

SUMMARY:
To monitor the quality of health care systems, patient-reported outcome measures (PROMs) should be collected and analyzed before and after medical interventions. The development of information technology and software along with an exponential increase in the use of the Internet now allows new modalities for collecting PROMs. Online survey has become one of the most popular methods of data collection. tHE hypothesis is that providing a "brace cold therapy" to patients undergoing knees surgeries will generate an increasing in Response Rate to Online surveys.

DETAILED DESCRIPTION:
In the setting of anterior cruciate ligament reconstruction (ACLR), an alternative to standard clinic-based follow-up is used in our institution via the utilization of Web-Based follow-up platform (OTHENSE) that allows surgeons to monitor a patient's subjective quality of recovery, including symptoms of pain and limitations in activities of daily living. This tool has the potential to enhance quality of care by providing weekly updates about the patient's physical impairment. We started using it in 2018.

From a single orthopedic surgeon, a total of 100 patients who were planned to undergo an ACLR requiring formal post-operative follow-up were participated.

The process began upon preop consultation, where the patient is offered a description of the survey and asked to use a link allowing direct access to the Online Surveys (ORTHENSE Platform).

• Participants were divided in two groups :

* First group: patients operated for ACLR
* Second group: patients operated for ACLR, and received a "knee brace cold therapy" to use it in the post op recovery rehabilitation, sent to patient's home directly during pre-op phase.

A standardized follow-up protocol for both groups.

The surveys included questions related to rehabilitation and questions from standard patient-reported-outcome-measures PROMs. They were asked to complete the following surveys pre-operatively and post-operatively:

J -14 / J-7 / J -5/ J-2 / J+3 / J+7 / J+14 / J+21 / J+28 / J+35 / J+45

For both groups, data was collected for up to 6 weeks following Surgery (J+45), for a total of 11 surveys

ELIGIBILITY:
Inclusion Criteria:

* Patients performing knee surgeries (ACL)
* 6 Weeks minimum of F/U (J+45)
* In University Hospital Toulouse

Exclusion Criteria:

* F/U = 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated for ACLR between May 2020 and April 2021
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
percentage of change in the Online surveys Response Rate between two groups with or without knee brace cold therapy | 45 days
  percentage of Response rate to 11 surveys

CONTACTS AND LOCATIONS:
Overall Officials: Etienne CAVAIGNAC, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No